CLINICAL TRIAL: NCT05569395
Title: Effects of Neuromobilization on Stiffness of Median Nerve: Randomized Controlled Trial
Brief Title: Effects of Neuromobilization on Median Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Kubra Koce, Asst. Prof., Istinye University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 100
Record Dates: First submitted 2022-09-15; First posted 2022-10-06 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Median Nerve; Neuromobilization; Stiffness

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Median nerve neuro mobilization group
  Interventions: Other: Neuro mobilization
- Control Group (Sham Comparator): Sham median nerve neuro mobilization group
  Interventions: Other: Sham neuro mobilization

INTERVENTIONS:
Other: Neuro mobilization — For median nerve stretching, the participants' dominant forearms will be in the supination position while the shoulder will be depressed and abducted 90 degrees.
  In this position, while the participant's head is lateral flexed to the opposite side, the wrist and finger will be extended and median nerve stretching will be performed. After staying in this position for 30 seconds, the participants will relax by placing the wrist and head in the neutral position. Thus, a set for median nerve stretching will be completed. For median nerve gliding, the dominant side of the individuals' forearms will be in supination, while the shoulder will be placed in a depression and 90 degree abduction position. In this position, the participant will flex the wrist and fingers while lateral flexing the head to the opposite side, and extend the wrist and fingers while the head is lateral flexed to the same side.
  Arms: Study group
Other: Sham neuro mobilization — Sham neuromobilization will be applied to the nondominant side upper extremities of the participants.
  Arms: Control Group

SUMMARY:
The median nerve is a mixed nerve with motor and sensory functions in the upper extremity. It is observed that the median nerve slides longitudinally during upper extremity movements. However, in entrapment neuropathies (eg, Carpal Tunnel Syndrome), longitudinal displacement of the nerve is partially limited. In addition, the presence of adhesion, fibrosis, and possible scar tissue may cause difficulties for peripheral nerve adaptation in certain positions and movements. This, in turn, can result in the limitation of nerve trunk movements with respect to the surrounding tissues and a reduction in the normal shift of nerve fibers and fascicles relative to each other and to the connective tissues. Any pathology that reduces the normal stretch and slip of the medial nerve produces abnormal tension during extremity movement and the pressure on the nerve increases. This may cause symptoms such as paresthesia, weakness, and pain in the hand. With neuromobilization exercises, the tension and pressure on the median nerve are reduced and the nerve is prevented from being compressed in the carpal tunnel.

Neuromobilization is part of manual therapy and has been reported to be an effective practice for some conditions, including low back pain and carpal tunnel syndrome. The inclusion of neuromobilization in the treatment of patients with carpal tunnel syndrome, cervicobrachial pain, and lateral epicondylitis, in particular, has been associated with a reduction in the degree of pain and disability. Recently, neuromobilization techniques have started to be used in the treatment of nerve compression. These techniques consist of a series of therapeutic active and passive movements aimed at restoring the normal mechanical properties of the nerve during limb movements.

When the literature is examined, there are not many studies that objectively reveal the effects of neuromobilization techniques on nerve elasticity. Shear Wave Elastography is a method that quantitatively reveals the elasticity of tissues by measuring the speed of shear waves formed in the tissues through non-invasive high-frequency ultrasound waves. In recent studies, Shear Wave Elastography has shown promising results in demonstrating the elasticity of peripheral nerves.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-30 years
* Healthy individuals without any known systemic disease

Exclusion Criteria:

* Those who had an upper extremity such as bone-tendon-muscle operation in the last six months
* Those with a systemic disease such as rheumatoid arthritis, diabetes mellitus
* Those with any neuromuscular disease (such as Multiple sclerosis, myopathy)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Median Nerve Tension Test | 1 week
  The test is performed with the participant in supine position with shoulder depression and 90 degrees abduction and external rotation, elbow 90 degrees flexion, forearm in full supination, and wrist and fingers in full extension. Maintaining this position, the elbow is passively extended to test the tension of the median nerve. The test is stopped at the point where the patient feels pain and tension, and the angle formed at the elbow will be measured with a universal goniometer and recorded. The measurement will be repeated 3 times and the average value will be recorded.
Shear Wave Ultrasound Elastography | 1 week
  Nerve elasticity will be measured by measuring the speed of shear waves formed in the median nerve by means of high frequency ultrasound waves.

SECONDARY OUTCOMES:
Range of Motion | 1 week
  Wrist flexion and extension will be measured bilaterally with a universal goniometer.
Finger Grip Strength | 1 week
  Finger grip strength will be measured bilaterally with a pinchmeter.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)